CLINICAL TRIAL: NCT02961166
Title: Intravenous Immunoglobulin Therapy in ARDS Patients With Extracorporeal Membrane Oxygenation (ECMO) Therapy
Brief Title: Immunglobulin M Enriched Intra Venous Immunoglobulin (IVIG) Therapy in Adult Respiratory Distress Syndrom (ARDS) Patients
Acronym: IVIG
Status: Completed | Type: Observational
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Universität Tübingen (Other)
Responsible Party: Principal Investigator, PD Dr. Helene Haeberle, PD Dr. med. Helene Haeberle, University Hospital Tuebingen
Other Study IDs: University Hospital Tuebingen
Record Dates: First submitted 2016-05-08; First posted 2016-11-10 (Estimated); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Respiratory Distress Syndrome, Adult; Septic Shock
Keywords: IVIG; ARDS; ECMO
MeSH Terms: conditions — Respiratory Distress Syndrome; Shock, Septic | interventions — pentaglobulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IgM enriched Immunoglobulins: ARDS patients with septic shock requiring ECMO therapy were treated for 3 days by IgM-enriched Immunoglobulin
  Interventions: Drug: IgM enriched Immunoglobulins
- Control: ARDS patients with septic shock requiring ECMO therapy were NOT treated by IgM-enriched Immunoglobulin

INTERVENTIONS:
Drug: IgM enriched Immunoglobulins — Treatment for 3 days
  Other Names: Pentaglobin, Biotest Pharma GmbH Germany; Code 170a/90
  Groups: IgM enriched Immunoglobulins

SUMMARY:
57 patients with Adult Respiratory Distress Syndrome (ARDS) requiring Extracorporeal membrane oxygenation (ECMO) therapy were analyzed retrospectively. 28 patients had received immunglobulin M-enriched immunoglobulin therapy (IVIG); 29 patients did not receive IVIG therapy.

These patients were analyzed regarding length of stay in intensive care unit (LOS ICU), length of stay (LOS) in hospital and regarding mortality.

DETAILED DESCRIPTION:
57 patients with ARDS requiring ECMO therapy were analyzed retrospectively. 28 patients had received IgM-enriched immunoglobulin therapy (IVIG); 29 patients did not receive IVIG therapy.

Patient characteristics, like Acute Physiology And Chronic Health Evaluation (APACHE) and Sepsis-related organ failure assessment (SAPS) Score, preexisting diseases, origin of infection, duration of ECMO therapy were analyzed in these patients.

These patients were further analyzed regarding LOS ICU, LOS in hospital and regarding mortality.

ELIGIBILITY:
Inclusion Criteria:

* All data available
* ARDS with ECMO therapy

Exclusion Criteria:

* Data missing

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ARDS patients treated by ECMO in the anesthesiological ICU of University Hospital Tuebingen between january 2012 and december 2015
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2012-01; Primary Completion 2016-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Mortality | during ICU treatment, up to 28 days
  Death during ICU therapy

SECONDARY OUTCOMES:
lengh of stay (LOS ICU) | up to 60 days
  lengh of stay on ICU in days

CONTACTS AND LOCATIONS:
Overall Officials: Helene A Haeberle, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Prohaska S, Schirner A, Bashota A, Korner A, Blumenstock G, Haeberle HA. Intravenous immunoglobulin fails to improve ARDS in patients undergoing ECMO therapy. J Intensive Care. 2018 Feb 26;6:11. doi: 10.1186/s40560-018-0278-8. eCollection 2018. PMID 29497534